CLINICAL TRIAL: NCT05239325
Title: Step up to Health, Nigeria! Utilizing Information From Abuja's 2022 World Cancer Day Walk for Equity-based Cancer Prevention Interventions
Brief Title: Step up to Health, Nigeria! Impact of 2022 World Cancer Day Walk on Health Behaviors Among Nigerians
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: AshtaYoga, LLC (Industry)
Collaborators: Project PINKBLUE, Health and Psychological Trust Centre (Unknown); University Of Nigeria Teaching Hospital (Network); Vaughan A. Lewis Institute for Research and Innovation (Other); Columbia University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Nigeria World Cancer Walk 2022
Record Dates: First submitted 2022-02-03; First posted 2022-02-14 (Actual); Last update posted 2022-02-14 (Actual); Status verified 2022-02

CONDITIONS: Cancer Prevention
Keywords: Nigeria; Cancer Prevention; Cancer Screening; Physical Activity; Health Literacy; Health Behaviors
MeSH Terms: conditions — Motor Activity; Health Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Active Comparator): Participants having previously attended at least once in previous years the "World Cancer Day Walk" will be considered as the group exposed to the health education intervention (returning).
  Interventions: Behavioral: World Cancer Day Walk
- Control Group (No Intervention): The control/non-exposed group will be the participants who are attending the "World Cancer Day Walk" for the first time in 2022 (first timers) and have not yet received health education information.

INTERVENTIONS:
Behavioral: World Cancer Day Walk — Health literacy education (cancer prevention and healthy lifestyle) and free breast, prostate, cervical cancer screening
  Arms: Intervention Group

SUMMARY:
Cancer awareness is a critical element of cancer prevention and control. Creating public awareness on risk factors, preventative strategies, and the importance of early screening is the foundation upon which a cancer control program must be constructed. The purpose of this study is to describe the sociodemographic and risk factor distribution of the Abuja, Nigeria "World Cancer Day Walk" participants according to their motive for participating in the event (free cancer screening versus fun/activities), and secondarily, to investigate the impact of the event on educating attendees from the general population about cancer prevention and screening, in particular the importance of being physically active and maintaining a healthy body weight. Obesity is a known risk factor contributing to the development of cancer and NCD's.

DETAILED DESCRIPTION:
Cancer awareness is a critical element of cancer prevention and control. Creating public awareness on risk factors, preventative strategies, and the importance of early screening is the foundation upon which a cancer control program must be constructed. Ideally, efforts should include knowledge of the problem and its solutions, a group of people who respect and care for the populations they want to serve, and importantly, resources.

Nigeria is the most populous black nation in the world with a population of over 196 million, more than 500 ethnic groups, 380 languages, and a diverse range of cultural, traditional and religious beliefs. Nigeria constitutes approximately 20% of the population of Africa and slightly more than 50% of the West African population. Cancer is a critical public health problem in this population. Nigeria is a major contributor to the overall cancer burden on the continent with 72,000 cancer deaths in 2012 and 115,950 new cases of cancer and 70,327 cancer deaths in 2018. Nigerians also have one of the world's poorest 5-year cancer survival rates.

Breast cancer is the most frequently diagnosed cancer in Nigerian women and the leading cause of cancer death in Nigeria, with an estimated 26,310 new cases and 11,564 deaths in 2018 (44% death rate). Breast cancer incidence in this population historically has been low but is now increasing. By comparison, in the United States (population 329 million) there were 30,700 new breast cancer cases and 6,310 deaths in 2016. Another female cancer - cervical, is 99% preventable, however, it is the second leading cause of cancer death in Nigeria with over 26 deaths every day. By comparison, in the United States between 2013-2017, the average annual death rate of cervical cancer was 2.3% per 100,000 (age adjusted to the 2000 US standard population). Prostate cancer is the leading cause of cancer deaths in Nigerian men with 13,078 new cases (which is 29.1%) and 5,806 deaths in 2018. The age-standardized incidence rates (ASR) for prostate cancer was 32.8 new cases per 100,000 men and mortality rate was about 16.3 per 100,000 men in 2018. On a daily basis, at least 15 men die of prostate cancer in Nigeria. By comparison, in the United States prostate cancer death rates in men declined 52% from 1993 to 2017.

Strategies for prevention and early detection are imperative in the reduction of cancer death rates globally; awareness campaigns (such as the annual "World Cancer Day Walk" in Abuja) are critical to educate the general population on cancer risk factors, the benefits of screening and early detection, and to offer free cancer screening to all populations.

This study "Step up to Health, Nigeria! Impact of the 2022 World Cancer Day Walk on Health Behaviors Among Nigerians" will describe the sociodemographic and risk factor distribution of the Abuja, Nigeria "World Cancer Day Walk" participants according to their motive for participation, and secondarily, to investigate the impact of the event on educating attendees from the general population about cancer prevention and screening, in particular the importance of being physically active and maintaining a healthy body weight. Obesity is a known risk factor contributing to the development of cancer and NCD's.

The study will take place in Abuja, Nigeria on Feb 5, 2022 during the 8th Annual "World Cancer Day Walk" sponsored by Project PINK BLUE, a registered Nigerian nonprofit cancer organization, viz. Health & Psychological Trust Centre (CAC/IT/NO 73960).

The purpose of the "World Cancer Day Walk" is to create awareness and advocate for better cancer care for Nigerians. The event offers free breast, cervical, and prostate cancer screenings; heath education and information about cancer risk reduction; and group physical activities that include a 5km Walk, 10km Race, 20km Ride, 5km Skate, 50km Cycle, and Marathon.

On the day of the event, the in-field research team will distribute a voluntary, one-page questionnaire to the anticipated 5,000 event participants to ascertain demographic information, cancer risk factors, motivations for attending the event, and lifestyle behaviors. Subjects will be recruited voluntarily onsite during the event following inclusion and exclusion criteria. Informed consent will be taken.

The questionnaire is 27 questions. Part one (eight questions) captures basic demographic information. Part two (six questions) captures personal and family history of cancer and cancer screening. Part three (six questions) captures information about the motivation for attending the event (free screening vs. fun/activities) and preferred ways to receive healthy lifestyle and cancer risk reduction / prevention information. Part four (five questions) captures lifestyle behaviors. Part five is the validated seven question International Physical Activity Questionnaire (IPAQ) instrument that measures physical activity and reduced sedentary behavior over the last seven days.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female age 18 and over
* Willing and able to converse and/or read and write in either English or Pidgin English.

Exclusion Criteria:

* Participants who are unable to provide informed consent to the study due to cognitive or physical impairment, based on self-report.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 527 (Estimated)
Dates: Start 2022-02-05 (Estimated); Primary Completion 2022-02-05 (Estimated); Study Completion 2022-02-05 (Estimated)

PRIMARY OUTCOMES:
Compare the sociodemographic and risk factor distribution of the "World Cancer Day Walk" participants who are attending the event for "free breast, cervical or prostate screening" with participants who are attending for "fun and activities". | Pre-intervention
  The brief survey instrument captures participant sociodemographic characteristics. Participants are asked to provide known risk factors for cancer and to indicate if they are attending for "free cancer screening" or "fun/activities".

SECONDARY OUTCOMES:
Compare physical activity metrics between those who are attending "World Cancer Day Walk" for the first time versus participants who have attended a previous "World Cancer Day Walk". | Pre-intervention
  The International Physical Activity Questionnaire (IPAQ) measures self-reported time spent per week doing vigorous and moderate activity in the last 7 days; time spent walking in the last 7 days, and time spent sitting down in the last 7 days. It is a "fill in the blank" survey instrument.

CONTACTS AND LOCATIONS:
Overall Officials: Leigh Leibel, MSc, Principal Investigator — Columbia University
Locations (1):
- Project Pink Blue, Abuja, Nigeria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rimer BK, Glassman B. Is there a use for tailored print communications in cancer risk communication? J Natl Cancer Inst Monogr. 1999;(25):140-8. doi: 10.1093/oxfordjournals.jncimonographs.a024190. PMID 10854470
- [Background] Oyetunde MO. Perception and management of cancer among the Yoruba in Ibadan, Nigeria. Afr J Med Med Sci. 2010 Sep;39(3):181-92. PMID 21416787
- [Result] Jemal A, Brawley OW. Increasing cancer awareness and prevention in Africa. Ecancermedicalscience. 2019 Jul 25;13:939. doi: 10.3332/ecancer.2019.939. eCollection 2019. PMID 31552112
- [Result] Jedy-Agba EE, Oga EA, Odutola M, Abdullahi YM, Popoola A, Achara P, Afolayan E, Banjo AA, Ekanem IO, Erinomo O, Ezeome E, Igbinoba F, Obiorah C, Ogunbiyi O, Omonisi A, Osime C, Ukah C, Osinubi P, Hassan R, Blattner W, Dakum P, Adebamowo CA. Developing National Cancer Registration in Developing Countries - Case Study of the Nigerian National System of Cancer Registries. Front Public Health. 2015 Jul 30;3:186. doi: 10.3389/fpubh.2015.00186. eCollection 2015. PMID 26284233
- [Result] Brawley OW. The role of government and regulation in cancer prevention. Lancet Oncol. 2017 Aug;18(8):e483-e493. doi: 10.1016/S1470-2045(17)30374-1. Epub 2017 Jul 26. PMID 28759387